CLINICAL TRIAL: NCT06718439
Title: Threshold for Operative and Postoperative Hemoglobin Trigger for Red Blood Cell Transfusion: A Pilot Randomized Controlled Trial (TOPGUN-Pilot)
Brief Title: Hemoglobin Levels for Blood Transfusions During and After Surgery
Acronym: TOPGUN-Pilot
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ottawa Hospital Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 20240690-01H
Record Dates: First submitted 2024-11-25; First posted 2024-12-05 (Actual); Last update posted 2025-07-31 (Actual); Status verified 2025-07

CONDITIONS: Blood Transfusion; Surgery
Keywords: Red blood cell transfusion; hemoglobin threshold; blood loss management; liberal transfusion practice; restrictive transfusion practice; intraoperative

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Restrictive transfusion strategy (Experimental): The restrictive transfusion strategy will consist of administering red blood cell transfusion when the participant's hemoglobin level is measured below 70 g/L or to maintain a hemoglobin target range of 70-80 g/L.
  Interventions: Procedure: Restrictive Transfusion
- Liberal transfusion strategy (Experimental): The liberal transfusion strategy will consist of administering red blood cell transfusion when the participant's hemoglobin level is measured below 90 g/L or to maintain a hemoglobin target range of 90-100 g/L.
  Interventions: Procedure: Liberal transfusion

INTERVENTIONS:
Procedure: Restrictive Transfusion — Red blood cell transfusion when the participant's hemoglobin level is measured below 70 g/L or to maintain a hemoglobin target range of 70-80 g/L. This strategy will be adhered to during surgery and up to 6 hours in the post-operative anesthesia care unit.
  Arms: Restrictive transfusion strategy
Procedure: Liberal transfusion — Red blood cell transfusion when the participant's hemoglobin level is measured below 90 g/L or to maintain a hemoglobin target range of 90-100 g/L. This strategy will be adhered to during surgery and up to 6 hours in the post-operative anesthesia care unit.
  Arms: Liberal transfusion strategy

SUMMARY:
The goal of this pilot clinical trial is to learn if it is achievable to conduct a large-scale clinical trial whereby, the investigators will compare two ways of deciding when to give a blood transfusion during surgery. Participants in this study are adults undergoing surgery with a risk of significant blood loss.

The main question it aims to answer is:

* Is a trial designed to definitively test and compare two different red blood cell transfusion strategies feasible?

Participants will:

* Receive blood transfusions during surgery based on a higher (less than 90 g/L) or a lower (less than 70 g/L) hemoglobin value.
* Complete questionnaires at 30 and 90 days after surgery.

DETAILED DESCRIPTION:
During some surgeries, there is a risk of significant blood loss. To manage this, blood transfusions may be needed to replace lost blood.

Transfusion strategies during surgery vary among physicians and hospitals. Current guidelines are broad and suggest it is okay to limit blood transfusions during surgery. However, some anesthesiologists worry that not giving enough blood might cause problems for patients. On the other hand, many cancer surgeons are concerned that giving too much blood could lead to worse outcomes for cancer patients. This difference in opinions shows why clinical trials are needed to guide future practices.

The purpose of this study is to test a new protocol that is designed to definitively test and compare two different red blood cell transfusion strategies. It is hypothesized that this trial will be deemed feasible.

TOPGUN-Pilot is a pragmatic, individually randomized, parallel-arm, vanguard, randomized controlled trial. If feasibility is demonstrated, patients enrolled in the vanguard pilot will be rolled into the definitive TOPGUN trial. This trial is meant to be pragmatic in nature, whereby the study protocol is simple to implement, outcomes are relevant to patients, physicians, and healthcare administrators, and data collection is limited. Management of patients prior to, during, and after the intraoperative transfusion strategies will be at the discretion of individual practitioners. A total of 384 patients will be randomized across 3 hospitals (4 sites) in Ontario and Quebec.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients, age ≥18.
* Elective or urgent surgery.
* Risk of red blood cell transfusion of at least 10 percent.
* Preoperative hemoglobin of less than 130 g/L.
* Intraoperative hemoglobin of ≤ 100 g/L at any time during surgery.

Exclusion Criteria:

* Active major hemorrhage as indication for surgery (e.g. ruptured aneurysm, polytrauma, etc.).
* Acute coronary syndrome or myocardial infarction within the past 6 weeks.
* Cardiac surgery.
* Liver transplantation.
* Surgery for moderate to severe (Glasgow Coma Scale (GCS) score ≤ 12) traumatic brain injury.
* Pregnancy or obstetrical surgery.
* Patient refusal of blood products.
* Inability to provide consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 384 (Estimated)
Dates: Start 2025-04-16 (Actual); Primary Completion 2026-04-15 (Estimated); Study Completion 2027-01-15 (Estimated)

PRIMARY OUTCOMES:
Recruitment rate | 12 months post site initiation
  Recruitment of ≥8 patients per month per site for one year.
Intervention adherence | From enrollment up to 6 hours in the Post-Anesthetic Care Unit
  Intervention adherence of at least 85%.
Participant retention | From randomization to 30 days post surgery.
  Retention of at least 90% of participants with completion of 30-day effectiveness outcomes.

CONTACTS AND LOCATIONS:
Overall Officials: Guillaume Martel, MD, MSc, FRCSC, FACS, Principal Investigator — Ottawa Hospital Research Institute
Locations (1):
- The Ottawa Hospital, Ottawa, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Undecided